CLINICAL TRIAL: NCT00362076
Title: Categorization Based on Motion-Carried Information in Infancy
Brief Title: The Role of Motion in Infants' Ability to Categorize
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980155; 98-CH-0155
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-04-19

CONDITIONS: Child Development
Keywords: Perception; Development; Cognition; Vision; Infants; Autonomic Function; Cardiac Vagal Tone; Categorization; Habituation; Motion-Carried Information
MeSH Terms: conditions — Substance-Related Disorders

SUMMARY:
This study is concerned with psychological and physiological development in infants. Specifically, researchers are interested in when and how babies are able to group similar objects, like animals or vehicles, into the same category. This study will investigate whether motion aids in the categorization process and allows for earlier demonstration of this competency.

Previous studies have demonstrated that the ability to categorize stationary objects or images of objects, is present by 6 months of age. This study is made up of three experiments to test:

1. The infant's ability to categorize photographic stimuli.
2. The infant's ability to categorize moving stimuli.
3. The infant's ability to transfer knowledge from moving to photographic stimuli.

Initially, the abilities of 3- and 6-month-old infants will be compared. It is also possible that 9-month-old infants will be tested. Data will consist of looking at time measures (level of attention to displays) and heart rate. The ability of infants to transfer category knowledge will support the view that motion is a source of information for object categorization.

DETAILED DESCRIPTION:
The major objective of this research is to better understand the early development of perceptual categorization. The proposed work is designed to examine the emergence of infants' ability to access internal categorical representations. Representation refers simply to stored information that can influence later behavior. Categorization refers to the treatment of discriminable objects as equivalent in some way. Even very young infants appear able to visually categorize diverse sets of discriminable patterns or objects. Much less is known, however, about how infants internally represent and utilize such information. The present set of studies is designed to probe the ontogeny of category of representations in infancy. The methodological strategy to be used in the first study consists of exposing infants to entirely novel configurations of objects for fixed amounts of time and later analyzing infants' examination and manipulation of those objects once they have become familiar. Infants will be exposed to these novel categories of objects at home over a 2-month period. Later, in a laboratory procedure, 5-month-old infants will be tested both with the familiar objects and similar test objects. A second study will utilize eye-tracking technology to examine the nature of infants' eye movements as they visually encode the individual members of complex categories such as animals and vehicles. Finally, a third study is being conducted to examine the relation between individual differences in infants' category learning and subsequent variability in language learning later on in childhood.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA

Infants will be selected for inclusion in Studies 1 and 2 on the basis of age, gestational status (i.e., term vs. preterm birth), visual normality, and general health status.

The initial group will be recruited to participate within two weeks of becoming 2 months of age.

Infants with a gestational age of less than 36 weeks, and/or those with histories of severe perinatal complications, visual abnormalities, or congenital developmental disorders will not be recruited for participation.

Equal numbers of males and females will be recruited to participate.

Ages: 3 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 941 (Actual)
Dates: Start 1998-09-03; Study Completion 2012-04-19

CONTACTS AND LOCATIONS:
Overall Officials: Jack A Yanovski, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Arterberry ME, Yonas A. Infants' sensitivity to kinetic information for three-dimensional object shape. Percept Psychophys. 1988 Jul;44(1):1-6. doi: 10.3758/bf03207466. No abstract available. PMID 3405724
- [Background] Bornstein MH, Kessen W, Weiskopf S. Color vision and hue categorization in young human infants. J Exp Psychol Hum Percept Perform. 1976 Feb;2(1):115-29. doi: 10.1037//0096-1523.2.1.115. PMID 1262792
- [Background] Behl-Chadha G. Basic-level and superordinate-like categorical representations in early infancy. Cognition. 1996 Aug;60(2):105-41. doi: 10.1016/0010-0277(96)00706-8. PMID 8811742